CLINICAL TRIAL: NCT02061267
Title: OLIVE OIL ON NAMPT AND ITS RELATION WITH POSTPRANDIAL INFLAMMATION AND ATHEROSCLEROSIS IN THE SETTING OF METABOLIC SYNDROME. The OLNAMS Project
Brief Title: Olive Oil and Nampt on Postprandial Inflammation and Atherosclerosis in the Setting of Metabolic Syndrome
Acronym: OLNAMS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Research Council, Spain (Other Government)
Responsible Party: Principal Investigator, Francisco Jose Garcia Muriana, Scientific Research Francisco Jose Garcia Muriana, National Research Council, Spain
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: AGL2011-29008
Record Dates: First submitted 2014-02-05; First posted 2014-02-12 (Estimated); Last update posted 2019-03-13 (Actual); Status verified 2019-03

CONDITIONS: Metabolic Syndrome
Keywords: Metabolic Syndrome; Olive Oil; Niacin
MeSH Terms: conditions — Metabolic Syndrome | interventions — Niacin; Butter; Fatty Acids; Olive Oil; Oleic Acid; Fish Oils; Docosahexaenoic Acids

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Niacin Control (Experimental): The subjects will receive a vitamin B3 supplement (2 g)
  Interventions: Dietary Supplement: Niacin
- Niacin + SAT (Experimental): The subjects will receive a vitamin B3 supplement (2 g) and a test meal with high-fat (containing 72% saturated fat, 22% carbohydrate, and 6% protein)
  Interventions: Dietary Supplement: Niacin; Dietary Supplement: Saturated meal
- Niacin + ROO (Experimental): The subjects will receive a vitamin B3 supplement (2 g) and a test meal with high-fat (containing 72% monounsaturated fat, 22% carbohydrate, and 6% protein)
  Interventions: Dietary Supplement: Niacin; Dietary Supplement: Monounsaturated meal
- Niacin + O3 (Experimental): The subjects will receive a vitamin B3 supplement (2 g) and a test meal with high-fat (containing 72% polyunsaturated omega-3 fat, 22% carbohydrate, and 6% protein)
  Interventions: Dietary Supplement: Niacin; Dietary Supplement: Polyunsaturated meal

INTERVENTIONS:
Dietary Supplement: Niacin — The subjects will receive a vitamin B3 supplement (2 g)
  Other Names: Vitamine B3; Nicotinic Acid
Dietary Supplement: Saturated meal — Test meal with high-fat (containing 72% saturated fat, 22% carbohydrate, and 6% protein)
  Other Names: Butter; Saturated fat
  Arms: Niacin + SAT
Dietary Supplement: Monounsaturated meal — Test meal with high-fat (containing 72% monounsaturated fat, 22% carbohydrate, and 6% protein)
  Other Names: Refined olive oil; olive oil; oleic acid
  Arms: Niacin + ROO
Dietary Supplement: Polyunsaturated meal — Test meal with high-fat (containing 72% polyunsaturated omega-3 fat, 22% carbohydrate, and 6% protein)
  Other Names: Fish oil; Omega-3; DHA; EPA
  Arms: Niacin + O3

SUMMARY:
The metabolic syndrome may be defined as the constellation of cardiovascular disease (CVD) risk factors that comprises obesity, type 2 diabetes, dyslipidemia, and hypertension. Lack of habitual physical activity and certain dietary patterns, including high-saturated fatty acids (SFA) intake, contribute to increase the risk of CVD, whereas the greatest risk reduction is related with monounsaturated fatty acids (MUFA), mainly from olive oil, and omega-3 polyunsaturated fatty acids (PUFA). Vitamin B3, as a major substrate for nicotinamide phosphoribosyltransferase (NAMPT), has also emerged as a nutritional intervention strategy for prevention of CVD.

NAMPT has been shown to exert activities of central importance to cellular energetics and innate immunity. Within the cell, NAMPT is the rate-limiting step in a salvage pathway of nicotinamide adenine dinucleotide (NAD+) biosynthesis. By virtue of this role, it can regulate cellular levels of NAD+ and thereby NAD+-consuming enzymes. NAMPT is also released by a variety of cells, and elevated levels can be found in the systemic circulation of subjects with a range of inflammatory disorders.

Recent evidences suggest that, primarily due to its high MUFA content, olive oil is useful as an optimal fat for the modulation of CVD risk factors in the postprandial state. In addition, NAMPT has been shown to correlate with triglycerides in the fasting plasma, and a potential regulatory role for fatty acids on NAMPT expression has been proposed.

The global aim of the project is to assess whether olive oil (MUFA), compared to other dietary fatty acids (SFA and omega-3 PUFA) and in association with vitamin B3 could have benefits on NAMPT-related inflammation and atherosclerosis. We hope to provide important novel insights on the relationship among dietary fatty acids, NAD+ metabolism, and metabolic syndrome. This aim is expected to be achieved in one principal objective:

To elucidate the influence of olive oil (MUFA), butter (SFA) or fish oil (omega-3 PUFA) meals supplemented by vitamin B3 on postprandial NAMPT modulation and its involvement on leukocyte inflammatory response in subjects with metabolic syndrome.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of metabolic syndrome

Exclusion Criteria:

* Subjects will be excluded if, allergic to dairy products, allergic to fish oil, vegetarian, tobacco smoker, current or recent (<4 wk) use of fish oil supplements or more than four times fish/week, received innoculations within 2 mo of starting the study or planned to during the study, donated or intended to donate blood from 2 mo before the study till 2 mo after the study, unstable body weight (no weight gain/loss >3 kg), medical condition that can interfere with the study outcome (i.e., biochemical evidence of active heart disease, renal impairment, hypothyroidism, liver dysfunction, etc.), use of medications know to interfere with glucose homeostasis or lipid metabolism, use of anti-inflammatory medication, hormone or cytokine or growth factor therapies, abuse of drugs and/or alcohol, participation in another biomedical study within 1 mo before the first screening visit, or not wanting to be informed about chance-findings during screening. Another exclusion criteria will be severe diabetes, which requires application of insuin and diabetes-related complications.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2012-01-01 (Actual); Primary Completion 2013-12 (Actual); Study Completion 2015-06-30 (Actual)

PRIMARY OUTCOMES:
Evolution of Metabolic parameters in postprandial state | t = 0, 2, 3, 4 and 6 hours
  Glucose, insulin, C-peptide, triglyceride, and NEFA levels in plasma will be measured at several time-points postprandially (t = 0, 2, 3, 4, and 6 h) using routine biochemical procedures. Different empiric indices of postprandial β-cell function and insulin sensitivity will be determined.
Evolution of Inflammatory markers in postprandial state | t = 0, 2, 3, 4 and 6 hours
  Inflammatory markers will be measured in plasma at several time-points postprandially (t = 0, 2, 3, 4, and 6 h) using appropriate methods (EIA, ELISA, and/or Bioplex multiplex system), and will include NAMPT, the acute phase protein (hsCRP), PAI-1, fibrinogen, transferrin, albumin, MPO (myeloperoxidase), and cytokines such as TNFα, IL-1β, IL-6, IL-8, IL-10, ICAM-1, MCP-1, leptin, and adiponectin, among other markers. For NAD+ content in plasma at fasting and postprandially, we will add 0.5 M ice-cold HClO4 to samples; after 2 min, we will collect 100 μL of supernatants by centrifugation at 3,000 g for 5 min, add 20 μL K2HPO4 (1 M) with cooling on ice and adjust pH to 7.2-7.4 with KOH. We will add 50 μL of supernatant to the reaction mixture containing 0.1 M sodiumpyrophosphate-semicarbazid (pH 8.8), absolute ethanol, and dH2O. We will assess NAD+ spectrophotometrically at 339 nm at 25 °C, as a mean difference in absorbance before and 6 min after addition of alcohol dehydrogenase.
Pharmacokinetic of Niacin and its metabolites | t = 0, 2, 3, 4 and 6 hours.
  Quantitation of nicotinic acid and its metabolites (nicotinamide, nicotinuric acid, and N-methyl-2-pyridone-5-carboxamide) will be assessed in postprandial plasma by LC-MS/MS.

CONTACTS AND LOCATIONS:
Overall Officials: Francisco José García Muriana, phD, Principal Investigator — National Research Counsil
Locations (1):
- Instituto de la Grasa, CSIC, Seville, Spain